CLINICAL TRIAL: NCT06745752
Title: Incidence, Severity, and Determinants of Upper Back, Lower Back, and Pelvic Girdle Pain in the Late Postpartum Period
Brief Title: Late Postpartum Period and Pain
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Sena Dilek Aksoy, Principal Investigator, Kocaeli University
Other Study IDs: sdilek12
Record Dates: First submitted 2024-12-13; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-04

CONDITIONS: Upper Back Pain; Lower Back Pain; Pelvic Girdle Pain
Keywords: postpartum period; upper back pain; lower back pain; pelvic girdle pain; incidence
MeSH Terms: conditions — Back Pain; Low Back Pain; Pelvic Girdle Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- postpartum women: In the study, the upper back, lower back and pelvic girdle pain status of the participants in the postpartum period will be monitored.

SUMMARY:
Upper back, lower back and pelvic girdle pain significantly affect women's lives, especially in the postpartum period. This study aimed to characterize the frequency and severity of upper back, lower back and pelvic girdle pain in the 0 to 2 months postpartum period. The study will be conducted as a cross-sectional and correlational study. Data will be collected using the Information Form and Brief Pain Inventory designed by the researchers. Data will be collected face to face with the participants at the end of the first week, the end of the first month and the end of the second month after birth. IBM SPSS Statistics 29.0 software will be used in the analysis of the data.

DETAILED DESCRIPTION:
Research questions

1. What are the prevalence rates of upper back, lower back, and pelvic girdle pain points during the 0-2 months postpartum period?
2. What are the severity rates of upper back, lower back, and pelvic girdle pain points during the 0-2 months postpartum period?
3. What are the determinants of upper back, lower back, and pelvic girdle pain points during the 0-2 months postpartum? The population of the study will consist of postpartum participants registered in a district family health center (FHC) in western Turkey, who meet the inclusion criteria and are willing to participate in the study. The total number of postpartum women registered in the family health center in the year before the study began was 383. Therefore, no sample calculation was made and all participants who gave birth within one year after the beginning of the study will be included in the study.

The data of the study will be collected using the Information Form, and Brief Pain Inventory.

Information Form: This form consists of 15 questions about sociodemographic and obstetric characteristics based on an extensive literature review on the topic.

Brief Pain Inventory: Developed by Cleeland and Ryan in 1994, the Pain Inventory consists of seven items related to pain intensity and the dimension of how pain interferes with daily activities.

Data collection The researcher will explain the purpose of the study to pregnant women who meet the inclusion criteria, invite them to participate, and obtain their consent. Data will be collected from participants at the end of the first postpartum week (when they attend the first postpartum follow-up visit and newborn heel prick test), at the end of the first month (day 28) (when they attend the second dose of neonatal hepatitis B vaccine), and at the end of the second month (week 8 postpartum) (when they attend the first dose of BCG, DTP-Hib-HBV, and IPV vaccines). At the first visit, participants will complete an information form and the Brief Pain Inventory. At the second and third meetings, they will complete only the Brief Pain Inventory.

Statistical analysis Statistical analysis will be performed using IBM SPSS Statistics 29.0 software (IBM Corp., Armonk, NY, USA). Sociodemographic data will be evaluated using descriptive statistical methods (frequency, percentage, mean, standard deviation). Kolmogorov-Smirnov test will be used as normality test. Independent samples analysis, correlation analysis and logistic regression analysis will be used in the analyses. Significance will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Participants who were 0-2 months postpartum,
* Could read and speak Turkish,
* Between the ages of 18-49.

Exclusion Criteria:

* Participants with past or current mental illness,
* Those taking antidepressant or anxiolytic medications,
* Rheumatoid arthritis,
* Ankylosing spondylitis,
* Scheuermann disease,
* Ehlers-danlos syndrome,
* Spinal surgery,
* Nerve root compression,
* Spondylolisthesis,
* Perineal edema,
* Hematoma,
* Wound dehiscence,
* Bladder catheterization,
* serious postpartum complications (internal bleeding, femoral artery embolism, pelvic fracture),
* Those whose babies are in the neonatal intensive care unit,
* Those who left the research unfinished.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Participants who had given birth, aged 18-49, were registered at a district family health center (FHC) in western Turkey, met the inclusion criteria, and volunteered to participate in the study.
Sampling Method: Probability Sample
Enrollment: 243 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of upper back pain, lower back pain, and pelvic girdle pain | Postpartum day 7.
  Filling out the tools used in the research (Information Form and Brief Pain Inventory)
Evaluation of upper back pain, lower back pain, and pelvic girdle pain | Postpartum day 28.
  Filling out the tools used in the research (Information Form and Brief Pain Inventory)
Evaluation of upper back pain, lower back pain, and pelvic girdle pain | Postpartum day 56.
  Filling out the tools used in the research (Information Form and Brief Pain Inventory)

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No